CLINICAL TRIAL: NCT04025905
Title: REMEDEMPLOI: Social Cognition Training and Vocational Rehabilitation
Brief Title: Social Cognition Training and Vocational Rehabilitation
Acronym: REMEDEMPLOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A00124-53
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Each participant is randomized in one of the two groups, defined by the type of treatment allocated: Social Cognition Training program or only Informations
Masking Description: Randomization will be stratified by site, and history of previous work in supported employment (≥ 1 year working in the ESAT prior to enrollment) so that each treatment is implemented in 3 groups of 10 people in each of the three centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Cognition Training Program (Experimental): This program is taken from two validated cognitive remediation programs: the SCIT program and the RC2S program : perception of social situations - emotional processes and social perception;interpretation of social situations - theory of mind and attributions;acting in social situations - social skills training
  Interventions: Behavioral: Social Cognition Training
- Informations program (Sham Comparator): Educational team Information will be given to participants about work environment, social environment, stress management, sleep management, treatments. It will also include socialization sessions with board games or cultural activities.
  Interventions: Behavioral: Informations

INTERVENTIONS:
Behavioral: Social Cognition Training — Evaluate the impact of the social cognition training on employment maintaining in transitional Workforce Assistance Facilities and Services.
  Arms: Social Cognition Training Program
Behavioral: Informations — informations about work environment, social environment, stress management, sleep management, treatments
  Arms: Informations program

SUMMARY:
Social cognition impairments, frequently encountered in Serial Mental Illness, reduce the ability to find and to keep a job. Cognitive remediation and social cognition training reduce the impact of cognitive impairments on work outcomes . The purpose of this research is to associate a social cognition training program to vocational rehabilitation in the transition network (transitional Workforce Assistance Facilities and Services) to help people to maintain their jobs and to access to work in an ordinary environment. To support the development of social cognition interventions, additional care (users will retain their usual medical follow-up) will be implemented within the Workforce Assistance Facilities and Services.

This project is part of a strong partnership between the Cognitive remediation network (health sector: rehabilitation centers) and the Transition network (medico-social sector: three Workforce Assistance Facilities and Services having partnerships with rehabilitation centers). This partnership has been experienced previously in the RemedRehab project funded by the 2012 hospital clinical research program (PHRC). This project was recently completed.

DETAILED DESCRIPTION:
Social cognition training concomitant to work help to maintain employment in transitional Workforce Assistance Facilities and Services .

Participation in the study will be offered to anyone with severe psychic disorders and a social cognition disorder who started working in one of the transitional Workforce Assistance Facilities and Services in the year prior to inclusion to limit selection bias.

The study population is defined by the transitional Workforce Assistance Facilities and Services users involved.

The diagnosis is not included in the inclusion criteria. It will, however, be established according to DSM-5 criteria for included users, who will benefit from a semi-structured interview .

The expected benefits in the social cognition training programgroup are: best job maintaining rate in transitional Workforce Assistance Facilities and Services , improvement of social cognition, improvement of interpersonal skills, improvement of self-esteem, improvement of professional insertion and improvement of the patient's vision of his place in society.

Participants enrolled in information group may expect benefits on socialization and empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a serious mental illness (The specific diagnosis is not included in the inclusion criteria. It will, however, be established according to DSM-5 criteria for included users, who will benefit from a semi-structured interview (MINI, Sheehan et al., 1998).
* Admission in an ESAT in the last year prior to enrollment
* Expected duration of employment beyond two years
* Tutor's agreement (for persons under tutorship)
* Affiliation to social insurance

Exclusion Criteria:

* Absence of a social cognition disorder at neuropsychological evaluations
* Simultaneous participation in a social cognition remediation program
* Insufficient level of understanding of French to participate in the group (verbal exchanges)
* Insufficient visual acuity to participate in the group (use of slideshow in the group sessions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total number of hours worked | 6 months
  Difference between the total number of hours worked compared to the number of working hours provided for in the work contract for 6 months

SECONDARY OUTCOMES:
Change from baseline in social cognitive | 6 months
  The Ambiguous Intentions Hostility Questionnaire (AIHQ): a measure for evaluating hostile social-cognitive biases in paranoia
Change from baseline in self-esteem | 6 months
  Self-Esteem Rating Scale - Short Form (SERS-SF). Self-esteem was assessed with the Self-Esteem Rating Scale-Short Form (SERS-SF) . The SERS is a 20-item self-rating scale with two subscales: positive and negative self-esteem.
Change from baseline in self-stigmatization | 6 months
  Internalized Stigma of Mental Illness scale (ISMI ). The ISMI scale was developed to measure the internalized stigma of people with a mental illness
Change from baseline in the recovery process | 6 months
  STages Of Recovery Instrument (STORI) The STORI consists of 50 items, presented in 10 groups of five. Each group represents one of the four process components of recovery: hope; identity; meaning; responsibility

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK NICOLAS, PhD, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No